CLINICAL TRIAL: NCT05671744
Title: Validation of a Cell-Based Technology for Non-Invasive-Prenatal-Diagnosis (CB-NIPD) Using Circulating Whole Fetal Cells From Maternal Peripheral Blood.
Brief Title: Fetal Cell Analysis From Maternal Blood
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Menarini Biomarkers Singapore (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: MBS21-CBNIPD-001
Record Dates: First submitted 2022-12-20; First posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-12

CONDITIONS: Prenatal Screening; Pregnancy Related; Genetic Disease
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood samples from pregnant women (Other): Samples of peripheral blood collected from pregnant women undergoing CVS or genetic amniocentesis
  Interventions: Other: Cell-based non-invasive prenatal testing

INTERVENTIONS:
Other: Cell-based non-invasive prenatal testing — Blood sampling

SUMMARY:
The aim of this clinical study is the evaluation of clinical performance of a cell-based non-invasive test technology for fetal aneuploidies and segmental imbalances detection in a high-risk pregnancies population.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a viable singleton or twin pregnancy
* Women who have already been selected by their treating physician to undergo an invasive fetal diagnostic procedure
* Participant is at least 18 years old and can provide informed consent

Exclusion Criteria:

* Unable to provide informed consent
* Prenatal diagnosis of clinical Chorioamnionitis
* Intake of drugs or exposure to teratogenic agents
* Infections that carry a risk of vertical transmission
* Known maternal viral diseases: HIV and HCV, HBV

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Fetal chromosomal abnormalities detection in circulating fetal cells, | 2 year
  Evaluation of clinical performance of a cell-based technology for fetal chromosomal abnormalities detection in circulating fetal cells, using maternal blood samples from a population of high-risk pregnancies undergoing clinically indicated fetal diagnostic procedures.

SECONDARY OUTCOMES:
Number of suitable fetal cells | 2 year
  Determination, for each participant sample, of the number of intact fetal cells recovered that are suitable for downstream analysis.
Fetal sex assessment | 2 year
  Early, non-invasive fetal sex assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda-Policlinico di Milano Ospedale Maggiore, Milan, Italy

IPD SHARING:
Plan to Share IPD: No